CLINICAL TRIAL: NCT03271697
Title: Efficacy Study of Astragalus Membranaceus on Aneurysmal Subarachnoid Hemorrhage
Brief Title: Astragalus Membranaceus on Aneurysmal Subarachnoid Hemorrhage
Acronym: AMASH
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chun-Chung Chen, Attending Surgeon, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH106-REC1-074
Record Dates: First submitted 2017-08-21; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Huang Qi; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AM group (Experimental): Treatment group will accept Astragalus Membranaceus(AM) t.i.w treatment for 14 days from second day of admission, in addition to standard ordinary treatment.
  Interventions: Drug: Astragalus Membranaceus
- Placebo group (Placebo Comparator): Control group will accept placebo t.i.w treatment for 14 days from the second day of admission, in addition to standard ordinary treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Astragalus Membranaceus — This research is trying to see if AM can enhance the clinical prognosis for spontaneous aneurysm ruptured subarachnoid hemorrhage patients.
  Other Names: Astragalus propinquus
  Arms: AM group
Drug: Placebo — as a comparator comparing with AM group
  Other Names: Starch
  Arms: Placebo group

SUMMARY:
This research is trying to see if AM can enhance the clinical prognosis for spontaneous aneurysm ruptured subarachnoid hemorrhage patients.

DETAILED DESCRIPTION:
Astragalus membranaceus (AM, Huang-Chi) is a Chinese herb used extensively in China as a traditional treatment to treat stroke for a long time, and a number of studies have shown that AM can reduce cerebral infarction area and has anti-oxidation activity. Our previous studies have demonstrated enhanced recovery of neurologic function in patients with acute hemorrhagic stroke who received AM. It is hypothesized that AM either reduces inflammatory response or reduces perihematomal edema.

Subarachnoid hemorrhage secondary to rupture of a cerebral aneurysm is a medical condition associated with a high morbidity and mortality; approximately 10-15% of patients die before reaching medical care, and overall mortality is approximately 45%. Of those that survive, 30% suffer permanent disability graded as moderate to severe, and two-thirds of survivors never return to the same quality of life as they had prior to their hemorrhage. A large number of patients (30-70%) who are able to make it to the hospital and have successful treatment of their aneurysm will develop delayed cerebral vasospasm that is related to the blood clot from their initial aneurysm rupture. Of patients that survive their initial aneurysm rupture, vasospasm results in an additional 7% mortality and another 7% of severe disabilities secondary to ischemic strokes from severe spasm of cerebral arteries.

This research is trying to see if AM can enhance the clinical prognosis for spontaneous aneurysm ruptured subarachnoid hemorrhage patients. All procedures done as a part of this study are standard hospital care procedures done to treat aneurysmal subarachnoid hemorrhage according to the AHA/ASA guideline.

ELIGIBILITY:
Inclusion Criteria:

* Patients who admitted to the hospital within 24 hours of onset of aneurysmal subarachnoid hemorrhage (SAH) stroke
* Subarachnoid hemorrhage documented on head CT
* Hunt Hess Grade 1-4
* Both Male and Female
* Age more than 20 and less than 80 years older
* Informed consent obtained from a patient or legal representative before enrollment

Exclusion Criteria:

* Traumatic or mycotic aneurysms
* Complication of serious heart or hepatic disease or infection or renal failure
* Malignant tumor
* Patients judged to be inappropriate by physician in charge
* Pregnant / breast feeding women
* Patients have enrolled or have not yet completed other investigational drug trials within 1 month before screening
* Ever stroke, and mRS≧3

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Clinical symptom | 90 days post discharge following AM treatment for aneurysmal subarachnoid hemorrhage
  evaluating recovery scale percentage at 90 days post discharge following AM treatment for aneurysmal subarachnoid hemorrhage

SECONDARY OUTCOMES:
IL-6 | 14 days post discharge following AM treatment for aneurysmal subarachnoid hemorrhage
  Interleukin 6, IL-6 in blood and cerebrospinal fluid
IL-1β | 14 days post discharge following AM treatment for aneurysmal subarachnoid hemorrhage
  Interleukin 1β, IL-1β in blood and cerebrospinal fluid
TNF-α | 14 days post discharge following AM treatment for aneurysmal subarachnoid hemorrhage
  Tumor Necrosis Factor-α, TNF-α in blood and cerebrospinal fluid
S100-β | 14 days post discharge following AM treatment for aneurysmal subarachnoid hemorrhage
  S100-β in blood and cerebrospinal fluid

IPD SHARING:
Plan to Share IPD: No